CLINICAL TRIAL: NCT04397263
Title: A Phase 3, Open-label, Multicenter Study to Evaluate the Safety and Efficacy of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease
Brief Title: A Study of Guselkumab in Participants With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR108801; CNTO1959CRD3003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease | interventions — guselkumab

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Guselkumab (Experimental): Participants will receive guselkumab by intravenous (IV) infusion, followed by guselkumab by subcutaneous (SC) injection. Participants who are eligible and willing to continue guselkumab may enter the Long-term extension (LTE) phase and continue to receive guselkumab.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered intravenously for the first 3 doses and then subcutaneously for the subsequent doses.
  Other Names: CNTO1959

SUMMARY:
The purpose of this study is to evaluate the safety of Guselkumab in participants with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Have Crohn's Disease (CD) or fistulizing CD of at least 3 months duration (defined as a minimum of 12 weeks), with colitis, ileitis, or ileocolitis, confirmed at any time in the past by radiography, histology, and/or endoscopy
* Have moderate to severe CD as assessed by CDAI components of stool frequency (SF), and abdominal pain (AP) scores, and endoscopic evidence
* Have screening laboratory test results within the protocol specified parameters
* A female participant of childbearing potential must have a negative urine pregnancy test result at screening and baseline
* Demonstrated intolerance or inadequate response to conventional or to biologic therapy for CD

Exclusion Criteria:

* Has complications of CD, such as symptomatic strictures or stenoses, short gut syndrome, or any other manifestation
* Unstable doses of concomitant Crohn's disease therapy
* Receipt of Crohn's disease approved biologic agents, investigational agents, or procedures outside of permitted time frame as specified in the protocol
* Prior exposure to p40 inhibitors or p19 inhibitors
* Any medical contraindications preventing study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2025-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (25):
- Japan (25):
  - KOKIKAI Tokatsu Tsujinaka Hospital, Abiko
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Hitachi General Hospital, Hitachi
  - Asahikawa Medical University Hospital, Hokkaido
  - Ofuna Chuo Hospital, Kamakura
  - Kishiwada Tokushukai Hospital, Kishiwada
  - Kumamoto University Hospital, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Kyorin University Hospital, Mitaka
  - Kenseikai Dongo Hospital, Nara
  - Hyogo Medical University Hospital, Nishinomiya Shi
  - Okayama University Hospital, Okayama
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Saga University Hospital, Saga
  - Kitasato University Hospital, Sagamihara
  - Saitama Medical Center, Saitama
  - Sapporo Tokushukai Hospital, Sapporo
  - Sendai Kosei Hospital, Sendai Miyagi
  - Jichi Medical University Hospital, Shimotsuke
  - National Center for Global Health and Medicine, Shinjuku
  - Tokyo Women's Medical University Hospital, Shinjuku-ku
  - Tokyo Metropolitan Bokutoh Hospital, Sumida Ku
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Toyama Prefectural Central Hospital, Toyama
  - National Hospital Organization Toyohashi Medical Center, Toyohashi

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Upon completion of the open-label treatment phase, participants were permitted to enter the long-term extension (LTE) phase. The LTE phase is ongoing and results will be published after the completion of the study.
Groups:
- Guselkumab 200 Milligrams (mg): Participants received guselkumab 200 mg by intravenous (IV) infusion induction doses at Weeks 0, 4, and 8, followed by guselkumab 200 mg subcutaneous (SC) injection maintenance doses at every 4 weeks (q4w) after Week 8 up to Week 44. The participants who were eligible and willing to continue guselkumab entered the Long-term extension (LTE) phase at Week 48 and continued to receive guselkumab 200 mg SC injection q4w from Week 48 in the LTE phase. A post treatment safety follow-up visit was conducted 12 weeks after last dose of study drug.
Period: Overall Study
Arm/Group | Guselkumab 200 Milligrams (mg)
Started | 38
Completed (Completed signified all participants who completed study Week 48 at clinical cutoff date (29-Feb-2024).) | 36
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 38
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Treatment-emergent AEs (TEAEs) were AEs with onset during the intervention phase or that were a consequence of a pre-existing condition that had worsened since baseline. All TEAEs including serious and non-serious AEs were reported.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 33

2. Primary Outcome: Number of Participants With Treatment-emergent Serious Adverse Events (TESAEs)
Description: Number of participants with TESAEs were reported. TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 3

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of Special Interest (TEAESI)
Description: Number of participants with TEAESI was reported. Active tuberculosis (TB) or malignancies were considered as TEAESIs. TEAESIs were AESIs with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 0

4. Primary Outcome: Number of Participants With Treatment-emergent Abnormalities in Hematology Laboratory Parameters
Description: Number of participants with treatment-emergent abnormalities in hematology laboratory parameters were reported. Laboratory tests included in hematology were hemoglobin, lymphocytes, neutrophils, platelet count, Total WBC (white blood cell) Count. National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) toxicity grades were Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Potentially Life-Threatening). TE abnormalities are laboratory abnormalities with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab. Here, "n"(number analyzed) signifies number of participants analyzed at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Hemoglobin (increased): Grade 1: number analyzed (Participants) | 37
  Hemoglobin (increased): Grade 1 | 0
  Hemoglobin (increased): Grade 2: number analyzed (Participants) | 37
  Hemoglobin (increased): Grade 2 | 0
  Hemoglobin (increased): Grade 3: number analyzed (Participants) | 37
  Hemoglobin (increased): Grade 3 | 0
  Hemoglobin (increased): Grade 4: number analyzed (Participants) | 37
  Hemoglobin (increased): Grade 4 | 0
  Hemoglobin (decreased): Grade 1: number analyzed (Participants) | 37
  Hemoglobin (decreased): Grade 1 | 18
  Hemoglobin (decreased): Grade 2: number analyzed (Participants) | 37
  Hemoglobin (decreased): Grade 2 | 2
  Hemoglobin (decreased): Grade 3: number analyzed (Participants) | 37
  Hemoglobin (decreased): Grade 3 | 3
  Hemoglobin (decreased): Grade 4: number analyzed (Participants) | 37
  Hemoglobin (decreased): Grade 4 | 0
  Lymphocytes (increased): Grade 1: number analyzed (Participants) | 37
  Lymphocytes (increased): Grade 1 | 0
  Lymphocytes (increased): Grade 2: number analyzed (Participants) | 37
  Lymphocytes (increased): Grade 2 | 0
  Lymphocytes (increased): Grade 3: number analyzed (Participants) | 37
  Lymphocytes (increased): Grade 3 | 0
  Lymphocytes (increased): Grade 4: number analyzed (Participants) | 37
  Lymphocytes (increased): Grade 4 | 0
  Lymphocytes (decreased): Grade 1: number analyzed (Participants) | 37
  Lymphocytes (decreased): Grade 1 | 5
  Lymphocytes (decreased): Grade 2: number analyzed (Participants) | 37
  Lymphocytes (decreased): Grade 2 | 7
  Lymphocytes (decreased): Grade 3: number analyzed (Participants) | 37
  Lymphocytes (decreased): Grade 3 | 4
  Lymphocytes (decreased): Grade 4: number analyzed (Participants) | 37
  Lymphocytes (decreased): Grade 4 | 0
  Neutrophils (decreased): Grade 1: number analyzed (Participants) | 37
  Neutrophils (decreased): Grade 1 | 7
  Neutrophils (decreased): Grade 2: number analyzed (Participants) | 37
  Neutrophils (decreased): Grade 2 | 7
  Neutrophils (decreased): Grade 3: number analyzed (Participants) | 37
  Neutrophils (decreased): Grade 3 | 0
  Neutrophils (decreased): Grade 4: number analyzed (Participants) | 37
  Neutrophils (decreased): Grade 4 | 0
  Platelets (decreased): Grade 1: number analyzed (Participants) | 37
  Platelets (decreased): Grade 1 | 1
  Platelets (decreased): Grade 2: number analyzed (Participants) | 37
  Platelets (decreased): Grade 2 | 0
  Platelets (decreased): Grade 3: number analyzed (Participants) | 37
  Platelets (decreased): Grade 3 | 0
  Platelets (decreased): Grade 4: number analyzed (Participants) | 37
  Platelets (decreased): Grade 4 | 0
  Total WBC Count (increased): Grade 1: number analyzed (Participants) | 37
  Total WBC Count (increased): Grade 1 | 0
  Total WBC Count (increased): Grade 2: number analyzed (Participants) | 37
  Total WBC Count (increased): Grade 2 | 0
  Total WBC Count (increased): Grade 3: number analyzed (Participants) | 37
  Total WBC Count (increased): Grade 3 | 0
  Total WBC Count (increased): Grade 4: number analyzed (Participants) | 37
  Total WBC Count (increased): Grade 4 | 0
  Total WBC Count (decreased): Grade 1: number analyzed (Participants) | 37
  Total WBC Count (decreased): Grade 1 | 9
  Total WBC Count (decreased): Grade 2: number analyzed (Participants) | 37
  Total WBC Count (decreased): Grade 2 | 9
  Total WBC Count (decreased): Grade 3: number analyzed (Participants) | 37
  Total WBC Count (decreased): Grade 3 | 0
  Total WBC Count (decreased): Grade 4: number analyzed (Participants) | 37
  Total WBC Count (decreased): Grade 4 | 0

5. Primary Outcome: Number of Participants With Treatment-emergent Abnormalities in Chemistry Laboratory Parameters
Description: Number of participants with treatment-emergent abnormalities in chemistry laboratory parameters were reported. Laboratory parameters included in clinical chemistry were albumin, corrected calcium, creatinine, glucose, potassium, sodium. NCI-CTCAE) toxicity grades were Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe), Grade 4 (Potentially Life-Threatening). TE abnormalities are laboratory abnormalities with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Albumin (decreased): Grade 1: number analyzed (Participants) | 37
  Albumin (decreased): Grade 1 | 0
  Albumin (decreased): Grade 2: number analyzed (Participants) | 37
  Albumin (decreased): Grade 2 | 1
  Albumin (decreased): Grade 3: number analyzed (Participants) | 37
  Albumin (decreased): Grade 3 | 0
  Albumin (decreased): Grade 4: number analyzed (Participants) | 37
  Albumin (decreased): Grade 4 | 0
  Corrected Calcium (increased): Grade 1: number analyzed (Participants) | 37
  Corrected Calcium (increased): Grade 1 | 0
  Corrected Calcium (increased): Grade 2: number analyzed (Participants) | 37
  Corrected Calcium (increased): Grade 2 | 0
  Corrected Calcium (increased): Grade 3: number analyzed (Participants) | 37
  Corrected Calcium (increased): Grade 3 | 0
  Corrected Calcium (increased): Grade 4: number analyzed (Participants) | 37
  Corrected Calcium (increased): Grade 4 | 0
  Corrected Calcium (decreased): Grade 1: number analyzed (Participants) | 37
  Corrected Calcium (decreased): Grade 1 | 3
  Corrected Calcium (decreased): Grade 2: number analyzed (Participants) | 37
  Corrected Calcium (decreased): Grade 2 | 0
  Corrected Calcium (decreased): Grade 3: number analyzed (Participants) | 37
  Corrected Calcium (decreased): Grade 3 | 0
  Corrected Calcium (decreased): Grade 4: number analyzed (Participants) | 37
  Corrected Calcium (decreased): Grade 4 | 0
  Creatinine (increased): Grade 1: number analyzed (Participants) | 37
  Creatinine (increased): Grade 1 | 2
  Creatinine (increased): Grade 2 | 1
  Creatinine (increased): Grade 3: number analyzed (Participants) | 37
  Creatinine (increased): Grade 3 | 0
  Creatinine (increased): Grade 4 | 0
  Glucose (decreased): Grade 1: number analyzed (Participants) | 37
  Glucose (decreased): Grade 1 | 1
  Glucose (decreased): Grade 2: number analyzed (Participants) | 37
  Glucose (decreased): Grade 2 | 1
  Glucose (decreased): Grade 3: number analyzed (Participants) | 37
  Glucose (decreased): Grade 3 | 0
  Glucose (decreased): Grade 4: number analyzed (Participants) | 37
  Glucose (decreased): Grade 4 | 0
  Potassium (increased): Grade 1: number analyzed (Participants) | 37
  Potassium (increased): Grade 1 | 0
  Potassium (increased): Grade 2: number analyzed (Participants) | 37
  Potassium (increased): Grade 2 | 1
  Potassium (increased): Grade 3: number analyzed (Participants) | 37
  Potassium (increased): Grade 3 | 0
  Potassium (increased): Grade 4: number analyzed (Participants) | 37
  Potassium (increased): Grade 4 | 0
  Potassium (decreased): Grade 1: number analyzed (Participants) | 37
  Potassium (decreased): Grade 1 | 0
  Potassium (decreased): Grade 2: number analyzed (Participants) | 37
  Potassium (decreased): Grade 2 | 5
  Potassium (decreased): Grade 3: number analyzed (Participants) | 37
  Potassium (decreased): Grade 3 | 0
  Potassium (decreased): Grade 4: number analyzed (Participants) | 37
  Potassium (decreased): Grade 4 | 0
  Sodium (increased): Grade 1: number analyzed (Participants) | 37
  Sodium (increased): Grade 1 | 0
  Sodium (increased): Grade 2: number analyzed (Participants) | 37
  Sodium (increased): Grade 2 | 0
  Sodium (increased): Grade 3: number analyzed (Participants) | 37
  Sodium (increased): Grade 3 | 0
  Sodium (increased): Grade 4: number analyzed (Participants) | 37
  Sodium (increased): Grade 4 | 0
  Sodium (decreased): Grade 1: number analyzed (Participants) | 37
  Sodium (decreased): Grade 1 | 0
  Sodium (decreased): Grade 2: number analyzed (Participants) | 37
  Sodium (decreased): Grade 2 | 0
  Sodium (decreased): Grade 3: number analyzed (Participants) | 37
  Sodium (decreased): Grade 3 | 0
  Sodium (decreased): Grade 4: number analyzed (Participants) | 37
  Sodium (decreased): Grade 4 | 0

6. Primary Outcome: Number of Participants With TEAEs of Infections
Description: Number of participants with TEAEs of infections were reported. TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 11

7. Primary Outcome: Number of Participants With TEAEs of Injection-site Reactions
Description: Number of participants with TEAEs of injection-site reactions were reported. A significant injection-site reaction was defined as an adverse reaction that was manifested through 1 or more of the following symptoms: significant bruising, erythema, hemorrhage, irritation, pain, pruritus at the site of injection. TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that has worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 3

8. Primary Outcome: Number of Participants With TEAEs Temporally Associated With Infusion
Description: Number of participants with TEAEs temporally associated with infusion were reported. TEAEs are AEs with onset during the intervention phase or that are a consequence of a preexisting condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 0

9. Primary Outcome: Number of Participants With TEAEs of Suicidal Ideation, Suicidal Behavior, or Self-Injurious Behavior Without Suicidal Intent
Description: TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline. The Columbia-suicide severity rating scale (C-SSRS) defined was 5 subtypes of suicidal ideation and 4 possible suicidal behaviors, as well as non-suicidal self-injurious behavior and completed suicide. The C-SSRS was an investigator-administered questionnaire: 1) No suicidal ideation or behaviors (including self-injurious behavior without suicidal intent): No further action was needed; 2) Suicidal ideation levels 1-3 or non-suicidal self-injurious behavior; participant risk is assessed by the investigator. 3) Suicidal ideation levels 4 or 5 or any suicidal behavior: participant risk assessed and referral to a mental health professional. If no events qualify for scores of 1 to 10, score of 0 was assigned (0= "no event that can be assessed on the basis of C-SSRS"). Higher scores indicated greater severity.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 0

10. Primary Outcome: Number of Participants With Clinically Significant Treatment-emergent Abnormalities in Vital Signs
Description: Number of participants with clinically significant treatment-emergent abnormalities in vital signs were reported. Vital signs included weight, pulse rate, temperature, respiratory rate, systolic blood pressure, and diastolic blood pressure. TEAEs are AEs with onset during the intervention phase or that are a consequence of a pre-existing condition that had worsened since baseline.
Time Frame: From baseline (Week 0) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 0

11. Primary Outcome: Number of Participants With Concomitant Medications for Crohn's Disease
Description: Number of participants with concomitant medications for Crohn's disease were reported.
Time Frame: From screening (Week -8) up to Week 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Oral amino salicylates | 28
  6- mercaptopurine/azathioprine | 16
  oral corticosteroids | 12

12. Secondary Outcome: Number of Participants With Clinical Response Through Week 48
Description: Number of participants with clinical response through Week 48 were reported. Clinical response was defined as a greater than or equal to (>=) 100-point reduction from baseline in CDAI score or CDAI score less than <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) in general: higher score indicated higher disease activities and a decrease in total CDAI score over time indicated improvement in disease activity.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: Full analysis set (FAS) included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Week 4 | 20
  Week 8 | 25
  Week 12 | 30
  Week 16 | 28
  Week 20 | 28
  Week 24 | 30
  Week 28 | 29
  Week 32 | 29
  Week 36 | 29
  Week 40 | 28
  Week 44 | 29
  Week 48 | 31

13. Secondary Outcome: Number of Participants With Clinical Remission Through Week 48
Description: Number of participants with clinical remission through Week 48 were reported. Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) in general: higher score indicated higher disease activities and a decrease in total CDAI score over time indicated improvement in disease activity.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Week 4 | 17
  Week 8 | 19
  Week 12 | 23
  Week 16 | 23
  Week 20 | 22
  Week 24 | 25
  Week 28 | 25
  Week 32 | 25
  Week 36 | 26
  Week 40 | 23
  Week 44 | 25
  Week 48 | 29

14. Secondary Outcome: Number of Participants With Patient-reported Outcome(s) (PRO)-2 Remission Through Week 48
Description: Number of participants with PRO-2 remission through Week 48 were reported. PRO-2 remission was defined as abdominal pain (AP) mean daily score at or below 1 and stool frequency (SF) mean daily score at or below 3, and no worsening of AP or SF from baseline. Mean daily AP score was defined as the sum of abdominal pain/cramps ratings in the previous 7 days in a diary card divided by the total number of days assessments were performed. Average daily SF score was defined as the sum of number of liquid or very soft stools in the previous 7 days in a diary card divided by the total number of days assessments were performed. Mean daily SF and AP scores score at a scheduled visit were not calculated if total number of days of assessment was less than 5. Higher PRO-2 scores indicated more severe disease.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants
  Week 4 | 6
  Week 8 | 12
  Week 12 | 16
  Week 16 | 16
  Week 20 | 19
  Week 24 | 18
  Week 28 | 21
  Week 32 | 19
  Week 36 | 20
  Week 40 | 21
  Week 44 | 23
  Week 48 | 22

15. Secondary Outcome: Change From Baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) Score at Week 48
Description: Change from baseline in SES-CD score at Week 48 were reported. The SES-CD score was used to evaluate endoscopic improvement. The SES-CD was based on the evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component was scored from 0 (best) to 3 (worst) for each segment, resulting in a total score of up to 15 for each component, except for the narrowing component which only attain a maximum total score of 11 because, the presence of a narrowing that cannot be passed can be only observed once. The total SES-CD score was the sum of all the component scores across all the segments and it ranged from 0 (best) to 56 (worst), where higher scores indicated more severe disease.
Time Frame: Baseline (Week 0) and Week 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
score on a scale | -6.4 (7.00)

16. Secondary Outcome: Serum Concentation of Guselkumab
Description: Serum concentration of guselkumab were reported.
Time Frame: Predose at Weeks 0, 4, 8, 12, 16, 20, 24, 32, 40, 48 and 1 hour post dose at Weeks 0, 4, 8
Population: Pharmacokinetics (PK) analysis set included all enrolled participants who received at least 1 complete dose of guselkumab and have at least 1 valid blood sample drawn for PK analysis after their first dose of guselkumab. Here, 'n' signifies the number of participants evaluable at each specified timepoint.
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (mcg/mL)
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
micrograms/milliliter (mcg/mL)
  Week 0: pre-dose | NA (NA) — NA signifies that mean were below the lowest quantification (BQL=0) and hence standard deviation (SD) was not calculated.
  Week 0: 1 hour post dose | 60.567 (7.8417)
  Week 4: pre-dose: number analyzed (Participants) | 36
  Week 4: pre-dose | 6.656 (2.5431)
  Week 4: 1 hour post dose: number analyzed (Participants) | 35
  Week 4: 1 hour post dose | 63.556 (10.7183)
  Week 8: pre-dose: number analyzed (Participants) | 35
  Week 8: pre-dose | 8.679 (3.1697)
  Week 8: 1 hour post dose: number analyzed (Participants) | 35
  Week 8: 1 hour post dose | 65.484 (7.8536)
  Week 12: pre-dose: number analyzed (Participants) | 35
  Week 12: pre-dose | 9.691 (4.4559)
  Week 16: pre-dose: number analyzed (Participants) | 35
  Week 16: pre-dose | 9.143 (4.3351)
  Week 20: pre-dose: number analyzed (Participants) | 35
  Week 20: pre-dose | 8.761 (4.3497)
  Week 24: pre-dose: number analyzed (Participants) | 35
  Week 24: pre-dose | 8.966 (4.6369)
  Week 32: pre-dose: number analyzed (Participants) | 34
  Week 32: pre-dose | 8.381 (3.7270)
  Week 40: pre-dose: number analyzed (Participants) | 34
  Week 40: pre-dose | 9.417 (5.3775)
  Week 48: pre-dose: number analyzed (Participants) | 33
  Week 48: pre-dose | 8.885 (4.4065)

17. Secondary Outcome: Number of Participants With Anti-Guselkumab Antibodies Through Week 48
Description: Number of participants with anti-guselkumab antibodies through Week 48 were reported.
Time Frame: From Week 0 through Week 48
Population: Immunogenicity analysis set included all enrolled participants who received at least 1 dose of guselkumab and had at least 1 observed post dose immune response data. Here, 'N' (number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 37
Participants | 1

18. Secondary Outcome: Number of Participants With Neutralizing-Guselkumab Antibodies Through Week 48
Description: Number of participants with neutralizing-guselkumab antibodies through Week 48 were reported.
Time Frame: From Week 0 through Week 48
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 1
Participants | 0

19. Secondary Outcome: Change From Baseline in Inflammatory Pharmacodynamic (PD) Marker: C-reactive Protein (CRP) Concentration
Description: Change from baseline in inflammatory PD marker of CRP concentration were reported.
Time Frame: Baseline (Week 0), Weeks 4, 8, 12, 16, 20, 24, 32, 40 and 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab. Here, 'n' signifies number of participants evaluable at each specified timepoints.
Measure: Median (Inter-Quartile Range); unit: milligrams per liter (mg/L)
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
milligrams per liter (mg/L)
  Week 4: number analyzed (Participants) | 37
  Week 4 | -1.65 [-38.90 to -0.15]
  Week 8: number analyzed (Participants) | 37
  Week 8 | -2.20 [-36.55 to -0.25]
  Week 12: number analyzed (Participants) | 37
  Week 12 | -2.40 [-44.20 to -0.20]
  Week 16: number analyzed (Participants) | 35
  Week 16 | -0.90 [-44.10 to -0.30]
  Week 20: number analyzed (Participants) | 35
  Week 20 | -0.70 [-45.20 to 0.20]
  Week 24: number analyzed (Participants) | 35
  Week 24 | -1.60 [-45.10 to -0.20]
  Week 32: number analyzed (Participants) | 34
  Week 32 | -1.25 [-30.50 to -0.40]
  Week 40: number analyzed (Participants) | 34
  Week 40 | -1.05 [-31.90 to -0.20]
  Week 48: number analyzed (Participants) | 34
  Week 48 | -1.65 [-33.40 to -0.10]

20. Secondary Outcome: Change From Baseline in Inflammatory PD Marker: Fecal Calprotectin (FC) Levels
Description: Change from baseline in inflammatory PD marker of FC levels were reported.
Time Frame: Baseline (Week 0), Weeks 4, 8, 12, 24, and 48
Population: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab. Here, 'n' signifies number of participants evaluable at each specified timepoint.
Measure: Median (Inter-Quartile Range); unit: milligrams per kilogram (mg/kg)
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
milligrams per kilogram (mg/kg)
  Week 4: number analyzed (Participants) | 36
  Week 4 | -270.0 [-817.0 to -45.0]
  Week 8: number analyzed (Participants) | 36
  Week 8 | -252.5 [-1614.5 to -79.0]
  Week 12: number analyzed (Participants) | 35
  Week 12 | -380.0 [-1563.0 to -110.0]
  Week 24: number analyzed (Participants) | 35
  Week 24 | -310.0 [-1722.0 to -87.0]
  Week 48: number analyzed (Participants) | 34
  Week 48 | -280.0 [-1678.0 to -123.0]

21. Secondary Outcome: Change From Baseline in Crohn's Disease Activity Index (CDAI) Score at Week 48 by Serum Guselkumab Concentration Quartiles at Week 48
Description: Change from baseline in CDAI score at Week 48 by serum guselkumab concentration quartiles at Week 48 were reported. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) in general: higher score indicated higher disease activities and a decrease in total CDAI score over time indicated improvement in disease activity.
Time Frame: At Week 48
Population: The PK/PD analysis set included all enrolled participants who had evaluable data of both PK and PD at the same visit which included Week 12, Week 24 or Week 48 visit. Here, 'N' (number of participants analyzed) signifies participants who were analyzed for this outcome measure and 'n' signifies number of participants evaluable at each specified concentration.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 33
score on a scale
  <= 1st Quartile Concentration: number analyzed (Participants) | 9
  <= 1st Quartile Concentration | -171.7 (152.12)
  > 1st Quartile and <= 2nd Quartile Concentration: number analyzed (Participants) | 8
  > 1st Quartile and <= 2nd Quartile Concentration | -137.6 (74.78)
  >2nd Quartile and <= 3rd Quartile Concentration: number analyzed (Participants) | 8
  >2nd Quartile and <= 3rd Quartile Concentration | -157.5 (124.85)
  > 3rd Quartile Concentration: number analyzed (Participants) | 8
  > 3rd Quartile Concentration | -146.0 (111.21)

22. Secondary Outcome: Number of Participants in Clinical Response at Week 48 by Serum Guselkumab Concentration Quartiles at Week 48
Description: Number of participants in clinical response at Week 48 by serum guselkumab concentration quartiles at Week 48 were reported. Clinical response was defined as a >=100-point reduction from baseline in CDAI score or CDAI score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) in general: higher score indicated higher disease activities and a decrease in total CDAI score over time indicated improvement in disease activity.
Time Frame: At Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 33
Participants
  <= 1st Quartile Concentration: number analyzed (Participants) | 9
  <= 1st Quartile Concentration | 8
  > 1st Quartile and <= 2nd Quartile Concentration: number analyzed (Participants) | 8
  > 1st Quartile and <= 2nd Quartile Concentration | 8
  >2nd Quartile and <= 3rd Quartile Concentration: number analyzed (Participants) | 8
  >2nd Quartile and <= 3rd Quartile Concentration | 7
  > 3rd Quartile Concentration: number analyzed (Participants) | 8
  > 3rd Quartile Concentration | 8

23. Secondary Outcome: Number of Participants in Clinical Remission at Week 48 by Serum Guselkumab Concentration Quartiles at Week 48
Description: Number of participants in clinical remission at Week 48 by serum guselkumab concentration quartiles at Week 48 were reported. Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score <150. The multi-item CDAI score assessed severity of illness by collecting information on 8 different Crohn's disease-related variables (extraintestinal manifestations, abdominal mass, weight, hematocrit, use of antidiarrheal drug(s) and/or opiates, total number of liquid or very soft stools, abdominal pain/cramps, and general well-being). The last 3 variables were scored over 7 days by the participant on a diary card. The total CDAI score ranged from 0 (improvement in disease activity) to 600 (more disease activity) in general: higher score indicated higher disease activities and a decrease in total CDAI score over time indicated improvement in disease activity.
Time Frame: At Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 33
Participants
  <= 1st Quartile Concentration: number analyzed (Participants) | 9
  <= 1st Quartile Concentration | 7
  > 1st Quartile and <= 2nd Quartile Concentration: number analyzed (Participants) | 8
  > 1st Quartile and <= 2nd Quartile Concentration | 7
  >2nd Quartile and <= 3rd Quartile Concentration: number analyzed (Participants) | 8
  >2nd Quartile and <= 3rd Quartile Concentration | 7
  > 3rd Quartile Concentration: number analyzed (Participants) | 8
  > 3rd Quartile Concentration | 8

24. Secondary Outcome: Number of Participants in Endoscopic Response at Week 48 by Serum Guselkumab Concentration Quartiles at Week 48
Description: Number of participants in endoscopic response at Week 48 by serum guselkumab concentration quartiles at Week 48 were reported. Endoscopic response was defined as >=50 % improvement from baseline in SES-CD score or SES-CD score less than or equal to (<=) 2. The SES-CD was based on evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component was scored from 0 (best) to 3 (worst) for each segment, resulting in a total score of up to 15 for each component, except for narrowing component which only attain a maximum total score of 11 because, presence of a narrowing that cannot be passed can be only observed once. The total SES-CD score was sum of all component scores across all segments and it ranged from 0 (best) to 56 (worst), where higher scores indicated more severe disease.
Time Frame: At Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 33
Participants
  <= 1st Quartile Concentration: number analyzed (Participants) | 9
  <= 1st Quartile Concentration | 4
  > 1st Quartile and <= 2nd Quartile Concentration: number analyzed (Participants) | 8
  > 1st Quartile and <= 2nd Quartile Concentration | 4
  >2nd Quartile and <= 3rd Quartile Concentration: number analyzed (Participants) | 8
  >2nd Quartile and <= 3rd Quartile Concentration | 5
  > 3rd Quartile Concentration: number analyzed (Participants) | 8
  > 3rd Quartile Concentration | 5

25. Secondary Outcome: Number of Participants in Endoscopic Remission at Week 48 by Serum Guselkumab Concentration Quartiles at Week 48
Description: Number of participants in endoscopic remission at Week 48 by serum guselkumab concentration quartiles at Week 48 were reported. Endoscopic remission: an SES-CD score <= 4 with at least a 2-point reduction from baseline and no sub score >1 in any individual subcomponent. The SES-CD was based on evaluation of 4 endoscopic components (presence/size of ulcers, proportion of mucosal surface covered by ulcers, proportion of mucosal surface affected by any other lesions, and presence/type of narrowing/strictures) across 5 ileocolonic segments. Each endoscopic component was scored from 0 (best) to 3 (worst) for each segment, resulting in total score of 15 for each component, except for narrowing component which only attain a maximum total score of 11 because, presence of a narrowing that cannot be passed can be only observed once. The total SES-CD score was sum of all component scores (all segments) & it ranged from 0 (best) to 56 (worst), where higher scores indicated more severe disease.
Time Frame: At Week 48
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 33
Participants
  <= 1st Quartile Concentration: number analyzed (Participants) | 9
  <= 1st Quartile Concentration | 2
  > 1st Quartile and <= 2nd Quartile Concentration: number analyzed (Participants) | 8
  > 1st Quartile and <= 2nd Quartile Concentration | 3
  >2nd Quartile and <= 3rd Quartile Concentration: number analyzed (Participants) | 8
  >2nd Quartile and <= 3rd Quartile Concentration | 4
  > 3rd Quartile Concentration: number analyzed (Participants) | 8
  > 3rd Quartile Concentration | 4

26. Secondary Outcome: Change From Baseline in the Average Daily Prednisone-equivalent (P.Eq) Oral Corticosteroid Dose (Excluding Budesonide) Through Week 48 Among Participants Receiving Oral Corticosteroids Other Than Budesonide at Baseline
Description: Change from baseline in the average daily P.Eq oral corticosteroid dose (excluding Budesonide) through Week 48 among participants receiving oral corticosteroids other than Budesonide at baseline were reported.
Time Frame: Baseline (Week 0), Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab. Here, 'N' (number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligram per day (mg/day)
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 4
milligram per day (mg/day)
  Week 4 | 0.00 (0.000)
  Week 8 | 0.00 (0.000)
  Week 12 | 0.00 (0.000)
  Week 16 | -9.06 (6.722)
  Week 20 | -13.13 (8.509)
  Week 24 | -13.75 (7.500)
  Week 28 | -13.75 (7.500)
  Week 32 | -13.75 (7.500)
  Week 36 | -13.75 (7.500)
  Week 40 | -13.75 (7.500)
  Week 44 | -13.75 (7.500)
  Week 48 | -13.75 (7.500)

27. Secondary Outcome: Number of Participants Not Receiving Concomitant Corticosteroids at Week 48 Among Participants Receiving Concomitant Corticosteroids at Baseline
Description: Number of participants not receiving concomitant corticosteroids at Week 48 among participants receiving concomitant corticosteroids at baseline were reported.
Time Frame: At Week 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 9

28. Secondary Outcome: Number of Participants Not Receiving Concomitant Corticosteroids for at Least 30 Days Prior to Week 48 Among Participants Receiving Concomitant Corticosteroids at Baseline
Description: Number of participants not receiving concomitant corticosteroids for at least 30 days prior to Week 48 among participants receiving concomitant corticosteroids at baseline were reported.
Time Frame: Up to Week 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 9

29. Secondary Outcome: Number of Participants Not Receiving Concomitant Corticosteroids for at Least 90 Days Prior to Week 48 Among Participants Receiving Concomitant Corticosteroids at Baseline
Description: Number of participants not receiving concomitant corticosteroids for at least 90 days prior to Week 48 among participants receiving concomitant corticosteroids at baseline were reported.
Time Frame: Up to Week 48
Population: The FAS included all enrolled participants who received at least 1 dose of guselkumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Guselkumab 200 Milligrams (mg)
Number analyzed (Participants) | 38
Participants | 9

ADVERSE EVENTS:
Time Frame: All cause mortality: From screening (Week -8) up to Week 48; SAEs and Other AEs: From baseline (Week 0) up to Week 48
Description: Safety analysis set included all enrolled participants who received at least 1 dose of guselkumab.
Arm/Group | Guselkumab 200 Milligrams (mg)
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 3/38
Other Adverse Events (participants affected / at risk) | 26/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Guselkumab 200 Milligrams (mg) (N=38)
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Guselkumab 200 Milligrams (mg) (N=38)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 2
Dental Caries (Gastrointestinal disorders) | 2
Injection Site Bruising (General disorders) | 2
Pyrexia (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 4
Tinea Pedis (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 6
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04397263/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT04397263/SAP_001.pdf